CLINICAL TRIAL: NCT02712203
Title: Measles-mumps-rubella and Measles-mumps-rubella-varicella Vaccines: Effect of Age at First Dose on Safety and Immunogenicity of the Measles Component.
Brief Title: MMR and MMRV Vaccines: Effect of Age at First Dose on Safety and Immunogenicity of the Measles Component.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Gaston De Serres, MD, PhD, CHU de Quebec-Universite Laval
Other Study IDs: 200783
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Measles
Keywords: Measles vaccine; Priorix; Priorix-Tetra; Age at vaccination
MeSH Terms: conditions — Measles | interventions — Measles-Mumps-Rubella Vaccine; measles, mumps, rubella, varicella vaccine; Priorix-Tetra vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 12 months: MMR vaccine / MMRV vaccine : administration of the first dose at 12 months of age
  Interventions: Biological: MMR vaccine / MMRV vaccine
- 13 months: MMR vaccine / MMRV vaccine : administration of the first dose at 13 months of age
  Interventions: Biological: MMR vaccine / MMRV vaccine
- 14 months: MMR vaccine / MMRV vaccine : administration of the first dose at 14 months of age
  Interventions: Biological: MMR vaccine / MMRV vaccine
- 15 months or more: MMR vaccine / MMRV vaccine : administration of the first dose at 12 months of age or older
  Interventions: Biological: MMR vaccine / MMRV vaccine

INTERVENTIONS:
Biological: MMR vaccine / MMRV vaccine — Subcutaneous injection, two doses
  Other Names: Priorix®; Priorix-Tetra®

SUMMARY:
Healthy children who received two doses of GlaxoSmithKline (GSK) Biologicals' live attenuated measles-mumps-rubella vaccine (MMR) or measles-mumps-rubella-varicella vaccine (MMRV) in their second year of life.The purpose of this study is to assess the effect of the age at administration of the first dose on the reactogenicity and immunogenicity of the measles component of these vaccines.

In addition, this study will evaluate if the effect of the age at first dose is modified by the type of vaccine administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject between 11 to 22 months at the time of first vaccination.
* Written informed consent obtained from the parent/guardian of the subject.

Exclusion Criteria:

* History of previous measles, mumps, rubella and/or varicella vaccination or disease or known exposure to any of these diseases within 30 days prior to the inclusion in the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, included the chronic administration (defined as more than 14 days) of immune-suppressants or other immune-modifying drugs within six months prior to the firs vaccine dose.
* History of any neurologic disorders or seizures.
* History of allergic diseases or reactions likely to be exacerbated by any component of the vaccines.
* Planned administration of a vaccine not foreseen by the study protocol from 30 days prior to each vaccination until 42-56 days after each vaccination

Ages: 11 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects aged 11 to 22 months selected to participate in clinical trials to assess the safety and immunogenicity of the GSK biological Priorix-Tetra™ in Germany, Austria, Finland, Greece, Poland, Czech Republic, Italy, Lithuania, Norway, Romania, Russian Federation, Slovakia, Sweden, United States and Puerto Rico.
Sampling Method: Non-Probability Sample
Enrollment: 5808 (Actual)
Dates: Start 2004-07; Primary Completion 2010-07 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Short term seropositivity rates & anti-measles antibody titers after vaccination with MMR or MMRV | At day 42 after administration of a dose of MMR or MMRV vaccine
  Antibody titers are expressed as Geometric Mean Concentrations (GMC) in mIU/mL. The cut-off for seropositivity is anti-measles antibody titer ≥ 150 mIU/mL (performed on seronegative subjects prior to vaccination).

SECONDARY OUTCOMES:
Injection site reaction | Days 0-3 after vaccination
  Injection site reaction is defined by the presence of pain, redness and swelling
Systemic symptoms | Days 0 - 42 after administration of a dose of MMR or MMRV vaccine
  Will include fever (defined as rectal temperature ≥38°C), general malaise and measles-like rash
Long term seropositivity rates and anti-measles antibody titers after vaccination with MMR or MMRV | 2 and 3 years after vaccination with 2 doses of MMR or MMRV vaccines
  Antibody titers are expressed as Geometric Mean Concentrations (GMC) in mIU/mL The cut-off for seropositivity is anti-measles antibody titer ≥ 150 mIU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Gaston De Serres, MD, PhD, Principal Investigator — CHU de Quebec-Universite Laval

REFERENCES:
- [Background] Czajka H, Schuster V, Zepp F, Esposito S, Douha M, Willems P. A combined measles, mumps, rubella and varicella vaccine (Priorix-Tetra): immunogenicity and safety profile. Vaccine. 2009 Nov 5;27(47):6504-11. doi: 10.1016/j.vaccine.2009.07.076. Epub 2009 Aug 7. PMID 19665608
- [Background] Schuster V, Otto W, Maurer L, Tcherepnine P, Pfletschinger U, Kindler K, Soemantri P, Walther U, Macholdt U, Douha M, Pierson P, Willems P. Immunogenicity and safety assessments after one and two doses of a refrigerator-stable tetravalent measles-mumps-rubella-varicella vaccine in healthy children during the second year of life. Pediatr Infect Dis J. 2008 Aug;27(8):724-30. doi: 10.1097/INF.0b013e318170bb22. PMID 18600190
- [Background] Knuf M, Habermehl P, Zepp F, Mannhardt W, Kuttnig M, Muttonen P, Prieler A, Maurer H, Bisanz H, Tornieporth N, Descamps D, Willems P. Immunogenicity and safety of two doses of tetravalent measles-mumps-rubella-varicella vaccine in healthy children. Pediatr Infect Dis J. 2006 Jan;25(1):12-8. doi: 10.1097/01.inf.0000195626.35239.58. PMID 16395096